CLINICAL TRIAL: NCT04449055
Title: A Pilot Study of Transcranial Magnetic Stimulation for Treatment of Methamphetamine Use Disorders
Brief Title: Pilot TMS for Methamphetamine Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ryan M. Carnahan (Other)
Collaborators: University of New Mexico (Other); University of Utah (Other)
Responsible Party: Sponsor-Investigator, Ryan M. Carnahan, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202001387
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Stimulant Dependence; Methamphetamine-dependence; Addiction, Drug
Keywords: methamphetamine; addiction treatment; transcranial magnetic stimulation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Randomized order of TMS site stimulated first
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- DPFC first (Experimental): Participants in this arm will undergo all study procedures including consent; pre-, during, and post-psychological assessments; pre- and post- MRI and fMRI; 16 treatments of dual target TMS over a 4-week period; and substance use-related assessments to include substance use, withdrawal symptoms, and cravings to use. This arm will receive the dorsolateral prefrontal cortex stimulation first.
  Interventions: Device: Transcranial Magnetic Stimulation--DPFC first, MPFC second
- MPFC first (Experimental): Participants in this arm will undergo all study procedures including consent; pre-, during, and post-psychological assessments; pre- and post- MRI and fMRI; 16 treatments of dual target TMS over a 4-week period; and substance use-related assessments to include substance use, withdrawal symptoms, and cravings to use. This arm will receive the medial prefrontal cortex stimulation first.
  Interventions: Device: Transcranial Magnetic Stimulation--MPFC first, DPFC second

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation--DPFC first, MPFC second — Participants will undergo 16 treatments consisting of intermittent theta burst stimulation targeting the dorsolateral prefrontal cortex and continuous theta burst stimulation targeting the medial prefrontal cortex, over a 4-week period that coincides with psychosocial treatment for methamphetamine use disorder. Both treatments will be delivered at each TMS treatment visit. The DPFC first group will receive stimulation to the dorsolateral prefrontal cortex first and medial prefrontal cortex second at each treatment visit.
  Other Names: Theta burst stimulation
  Arms: DPFC first
Device: Transcranial Magnetic Stimulation--MPFC first, DPFC second — Participants will undergo 16 treatments consisting of intermittent theta burst stimulation targeting the dorsolateral prefrontal cortex and continuous theta burst stimulation targeting the medial prefrontal cortex, over a 4-week period that coincides with psychosocial treatment for methamphetamine use disorder. Both treatments will be delivered at each TMS treatment visit. The MPFC first group will receive stimulation to the medial prefrontal cortex first and DPFC second at each treatment visit.
  Other Names: Theta burst stimulation
  Arms: MPFC first

SUMMARY:
This is a pilot study to test the feasibility of a recruitment strategy and study protocol to examine the effects of a dual target transcranial magnetic stimulation treatment in methamphetamine use disorder. The study will test intermittent theta burst stimulation (TBS) targeting the dorsolateral prefrontal cortex (DLPFC) combined with continuous TBS targeting the medial prefrontal cortex (MPFC) in people with methamphetamine use disorder (MAUD) who are engaged in psychosocial treatment. We will randomize the order in which these treatments are delivered at each treatment session, but all subjects will receive both treatments. Intermittent TBS targeting the DLPFC is approved by the Food and Drug Administration for major depressive disorder, and continuous TBS targeting the MPFC has been studied in cocaine use disorder. We will administer this dual target TBS daily for 2 weeks, followed by three times weekly for 2 weeks, and monitor depressive symptoms, anxiety, sleep, craving, quality of life, and methamphetamine use for three months. Changes in functional connectivity of brain circuits will be evaluated with functional magnetic resonance imaging (fMRI) before and after treatment. We expect to observe changes in connectivity between the DLPFC, MPFC, and other regions implicated in addiction and impulsivity. Furthermore, we will evaluate if baseline differences in functional connectivity can be used to predict response. Psychological tests focusing on state impulsivity and risk taking will be administered, and we expect to observe reductions in these characteristics after treatment. We will test this protocol in 20 patients recruited from clinical care settings at University of Iowa Hospitals and Clinics, University of New Mexico Health System, and University of Utah Health to illustrate the feasibility of recruitment and completing the protocol, to support an external funding proposal.

DETAILED DESCRIPTION:
Overview: This is a two-arm randomized controlled trial. Participants with MAUD will receive 16 sessions of dual-target theta burst stimulation to the DLPFC and MPFC over 4 weeks. Participants will be randomized to whether they receive stimulation to the DLPFC or MPFC first, but both sites will be stimulated at each treatment. We will follow outcomes for 12 weeks. Outcomes include treatment retention, craving, self-reported MA or stimulant use, urine drug screen results, depressive symptoms, anxiety symptoms, sleep quality, quality of life, response inhibition, and functional connectivity. Magnetic resonance imaging (MRI) to measure functional connectivity and a flanker task to measure response inhibition will be completed at baseline and four weeks. More detail is provided in the outcome measures section. Subjects will also complete the Big Five Inventory at baseline, a measure of personality characteristics, to explore how these relate to outcomes including retention in treatment and the study.

MR Image Acquisition: MRI will be completed at baseline and after the last TMS session. The MRI sessions will be conducted using research dedicated MRI scanners at each site. Anatomical images will include volumetric T1 and T2 weighted images with a 1.0 mm isotropic spatial resolution. Resting state fMRI will be performed to collect 20 minutes worth of data.

Statistical Analysis:

Retention in the Study and Psychosocial Treatment: We will describe the proportion of subjects who complete the 4-week TMS treatment period and complete each subsequent monthly follow-up visit, depending on randomization group. We will use Kaplan-Meier curves to describe retention in the study and in psychosocial treatment, and log-rank tests to compare them. If non-retention is common enough, we will use Cox regression to explore baseline measures as predictors of retention. We anticipate that multivariate analysis will not be feasible with the sample size.

Symptoms and Impulse Control Measures: Primary analyses for other measures will focus on changes over the 4-week TMS treatment period. Changes in symptoms evaluated weekly or biweekly (e.g. craving, depression, affect, anxiety, sleep) will be assessed using generalized linear mixed models with appropriate distributions. We anticipate a Poisson distribution for days of MA or other stimulant use and will use a binomial distribution with a logit link to evaluate changes in positive urine drug screens. Randomization group by time interactions will be the primary variables of interest to assess the differences between slopes of change between groups during treatment. Paired t-tests or Wilcoxon signed-rank tests will be used to evaluate changes in measures completed at baseline and after 4 weeks of treatment. We will compare measures at baseline and 4 weeks to those at 8 weeks and 12 weeks similarly, but in separate analyses since decay in effects may occur after TMS ends.

Functional Connectivity Analysis: fMRI functional connectivity analysis will be performed using a standard analysis pipeline. Functional images will undergo pre-processing including brain extraction, motion correction, spatial smoothing (6 mm FWHM), and temporal filtering (.008 Hz < f < 0.08 Hz). Following preprocessing, the fMRI signal will be corrected for potential sources of noise using image-based estimates and motion correction parameters. The resulting corrected time-series will be used for all functional connectivity analyses. Functional connectivity will be measured by extracting time-series data from the pre-processed imaging data for the regions of interest (ROIs). Multiple ROIs will be examined and will be defined as spheres (6mm radius) based on coordinate locations previously published by Yeo and colleagues. Specifically, we will focus on connectivity in the cingulo-opercular network involved in cognitive control and salience (DLPFC - anterior insula; DLPFC - anterior cingulate) and reward processing/motivation circuit (MPFC - ventral striatum). Analyses will be averaged across right and left hemispheres but we will also explore differences between right and left hemispheres. The time series from the ROIs will be cross-correlated with the time-series from the other ROIs to determine the strength of functional connectivity between regions. The resulting Pearson's r will be converted to Fisher's z scores to improve normality for the statistical analysis. We will treat each ROI pair connection (DLPFC - anterior insula, DLPFC - anterior cingulate, MPFC - ventral striatum) as a dependent variable. Primary analyses will use Wilcoxon rank-sum tests to compare changes in connectivity at baseline vs. after TMS treatment between groups. We will explore correlates of connectivity and changes using Pearson or Spearman correlations and linear regression or mixed models.

Exploratory Analysis: Follow-up exploratory voxel-wise analyses will be conducted for functional connectivity, which will provide thousands of individual predictors. This will help confirm findings in large parcel ROI based analysis. We will use the same statistical models as used for the ROI based analysis described above but at the voxel level. Voxel-wise data creates a high-dimensional problem in which the number of predictors far exceeds the number of participants. Machine learning methods, such as random forest will be used to handle the high-dimensional sub-analyses. Random forest requires a minimum of data assumptions, automatically accounts for non-linear and interaction effects, and it has proven useful in identifying useful predictors in high-dimensional contexts.

Comparison with Historical Controls: We will compare retention in psychosocial treatment programs and positive urine drug screens from chart review with between the two randomization groups. Treatment retention will be compared using a log-rank test. Positive urine drug screens in each week of follow-up will be compared using generalized estimating equation models with a logit link, clustered on subject, with participation in the TMS study as the variable of interest.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with an active methamphetamine use disorder
* Is engaged in psychosocial treatment or articulates a plan to engage in psychosocial treatment for methamphetamine use disorder during the study period
* Age 18 to 60 years
* Able to consent for treatment and research participation
* English-speaking
* Receiving care from UIHC's Addiction Medicine service. This includes patients in the Crisis Stabilization Unit, seen by the inpatient consultation service, enrolling in partial hospitalization or intensive outpatient treatment, or seen in the outpatient Addiction Medicine clinics.

Exclusion Criteria:

* Age less than 18 years
* Patients that are excluded during TMS assessment including: patients with epilepsy or seizure disorder, patients with implanted ferromagnetic equipment in their face or skull near the stimulation target.
* Current medical treatment with clozapine or stimulants.
* Current diagnosis of bipolar disorder, schizoaffective disorder, schizophrenia, that is deemed by research team psychiatrists not to have been drug-induced. Psychotic disorder not associated with drug use per the MINI International Neuropsychiatric Interview. Psychosis NOS, in remission, or drug-induced psychotic episodes are not exclusion criteria since these may be related to methamphetamine misuse.
* Lacks the mental capacity to provide informed consent (i.e. not able to demonstrate understanding of the risks and benefits of participation)
* Has a court appointed guardian.
* Unstable medical illness.
* Current diagnosis of neurological disorder or neurocognitive disorder.
* Prior neurosurgical procedure.
* History of seizure.
* History of ECT treatment within the past three months.
* History of any previous TMS treatment.
* Known inability to complete the protocol, as assessed by asking them if they are able to make it to all visits for this study without assistance.

MRI Exclusion criteria:

* Implanted device including pacemaker, coronary stent, defibrillator, or neurostimulation device that is not MRI-compatible
* Metal in body including bullets, shrapnel, metal slivers
* Claustrophobia
* Uncontrolled high blood pressure
* Atrial fibrillation
* Significant heart disease
* Hemodynamic instability
* Kidney disease
* Pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Carnahan, PharmD, MS, Principal Investigator — University of Iowa; Alison C Lynch, MD, MS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Courtney KE, Ray LA. Methamphetamine: an update on epidemiology, pharmacology, clinical phenomenology, and treatment literature. Drug Alcohol Depend. 2014 Oct 1;143:11-21. doi: 10.1016/j.drugalcdep.2014.08.003. Epub 2014 Aug 17. PMID 25176528
- [Background] Ma T, Sun Y, Ku Y. Effects of Non-invasive Brain Stimulation on Stimulant Craving in Users of Cocaine, Amphetamine, or Methamphetamine: A Systematic Review and Meta-Analysis. Front Neurosci. 2019 Oct 18;13:1095. doi: 10.3389/fnins.2019.01095. eCollection 2019. PMID 31680830
- [Background] Zhang JJQ, Fong KNK, Ouyang RG, Siu AMH, Kranz GS. Effects of repetitive transcranial magnetic stimulation (rTMS) on craving and substance consumption in patients with substance dependence: a systematic review and meta-analysis. Addiction. 2019 Dec;114(12):2137-2149. doi: 10.1111/add.14753. Epub 2019 Aug 16. PMID 31328353
- [Background] Makani R, Pradhan B, Shah U, Parikh T. Role of Repetitive Transcranial Magnetic Stimulation (rTMS) in Treatment of Addiction and Related Disorders: A Systematic Review. Curr Drug Abuse Rev. 2017;10(1):31-43. doi: 10.2174/1874473710666171129225914. PMID 29189190
- [Background] Liang Y, Wang L, Yuan TF. Targeting Withdrawal Symptoms in Men Addicted to Methamphetamine With Transcranial Magnetic Stimulation: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Nov 1;75(11):1199-1201. doi: 10.1001/jamapsychiatry.2018.2383. PMID 30208372

RESULTS

PARTICIPANT FLOW:
Groups:
- DPFC First: Participants in this arm will undergo all study procedures including consent; pre-, during, and post-psychological assessments; pre- and post- MRI and fMRI; 16 treatments of dual target TMS over a 4-week period; and substance use-related assessments to include substance use, withdrawal symptoms, and cravings to use. This arm will receive the dorsolateral prefrontal cortex stimulation first.
  Transcranial Magnetic Stimulation: Participants will undergo 16 treatments consisting of intermittent theta burst stimulation targeting the dorsolateral prefrontal cortex and continuous theta burst stimulation targeting the medial prefrontal cortex, over a 4-week period that coincides with psychosocial treatment for methamphetamine use disorder.
- MPFC First: Participants in this arm will undergo all study procedures including consent; pre-, during, and post-psychological assessments; pre- and post- MRI and fMRI; 16 treatments of dual target TMS over a 4-week period; and substance use-related assessments to include substance use, withdrawal symptoms, and cravings to use. This arm will receive the medial prefrontal cortex stimulation first.
  Transcranial Magnetic Stimulation: Participants will undergo 16 treatments consisting of intermittent theta burst stimulation targeting the dorsolateral prefrontal cortex and continuous theta burst stimulation targeting the medial prefrontal cortex, over a 4-week period that coincides with psychosocial treatment for methamphetamine use disorder.
Period: Overall Study
Arm/Group | DPFC First | MPFC First
Started | 6 | 5
Completed | 1 | 3
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Missed 4 treatments--removed by PI | 1 | 1
Not completed — Could not refrain from methamphetamine for 24 hours before treatment--removed by PI | 1 | 0
Not completed — Incarcerated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who were randomized and received at least one treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | DPFC First | MPFC First | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (10.9) | 39.6 (10.5) | 38.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Retention in the Study
Description: Time to study dropout (to assess feasibility and tolerability of the protocol)
Time Frame: Baseline to 12 weeks (continuous)
Population: Participants who received at least one treatment.
Measure: Mean (Standard Error); unit: Days
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Days | 28.2 (9.4) | 45.4 (13.4)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Log-rank test; Test type: Superiority; p = 0.1760, Log Rank; chi-square = 1.8311

2. Primary Outcome: Retention in Psychosocial Treatment
Description: Time to discontinuation of psychosocial treatment
Time Frame: Baseline to 18 days (continuous--assessed weekly)
Population: Those randomized with complete data on continuation of psychosocial treatment for methamphetamine use disorder. Missing data due to a collection form error led to no information after 18 days, and information was not entered for some participants at earlier visits.
Measure: Median (95% Confidence Interval); unit: Days until discontinuation
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 5 | 4
Days until discontinuation | NA [NA to NA] — Median survival times were not estimable due to too few events | NA [NA to NA] — Median survival times were not estimable due to too few events
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; The null hypothesis is that time to discontinuation of psychosocial treatment is not different between groups; Test type: Superiority; p = 0.3711, Log Rank; chi-square = 0.8000 — Median and mean survival times were not estimable due to the small number of dropouts. Thus, we reported the proportion remaining in treatment at 18 days as the descriptive summary measure
Statistical Analysis 2: Comparison: DPFC First vs MPFC First; This test compared time to discontinuation of psychosocial treatment between groups; Test type: Superiority; p = 0.3711, Log Rank; chi-square = 0.8000

3. Secondary Outcome: Functional Connectivity of the Dorsolateral Prefrontal Cortex and Anterior Insula
Description: Functional connectivity of the dorsolateral prefrontal cortex and anterior insula (mean of left and right side connectivity) measured with fMRI, as defined by the temporal correlation in the blood-oxygen-level-dependent signals of the regions. Higher correlations indicate stronger functional connectivity.
Time Frame: Baseline, 4 weeks
Population: Participants with MRI data for both baseline and after 4 weeks of treatment.
Measure: Mean (Standard Deviation); unit: Pearson correlation (r)
Groups:
- DPFC First: Participants in this arm will undergo all study procedures including consent; pre-, during, and post-psychological assessments; pre- and post- MRI and fMRI; 16 treatments of dual target TMS over a 4-week period; and substance use-related assessments to include substance use, withdrawal symptoms, and cravings to use. This arm will receive the dorsolateral prefrontal cortex stimulation first and medial prefrontal cortex stimulation second at each treatment visit.
  Transcranial Magnetic Stimulation: Participants will undergo 16 treatments consisting of intermittent theta burst stimulation targeting the dorsolateral prefrontal cortex and continuous theta burst stimulation targeting the medial prefrontal cortex, over a 4-week period that coincides with psychosocial treatment for methamphetamine use disorder.
- MPFC First: Participants in this arm will undergo all study procedures including consent; pre-, during, and post-psychological assessments; pre- and post- MRI and fMRI; 16 treatments of dual target TMS over a 4-week period; and substance use-related assessments to include substance use, withdrawal symptoms, and cravings to use. This arm will receive the medial prefrontal cortex stimulation first and dorsolateral prefrontal cortex stimulation second at each treatment visit.
  Transcranial Magnetic Stimulation: Participants will undergo 16 treatments consisting of intermittent theta burst stimulation targeting the dorsolateral prefrontal cortex and continuous theta burst stimulation targeting the medial prefrontal cortex, over a 4-week period that coincides with psychosocial treatment for methamphetamine use disorder.
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 2 | 4
Pearson correlation (r)
  Temporal correlation between regions at baseline | -0.0437533 (0.0404869) | 0.000470725 (0.1561368)
  Temporal correlation between regions after 4-week intervention | 0.0844848 (0.0315233) | 0.0129312 (0.0308713)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority — Exact Wilcoxon rank-sum test comparing changes in temporal correlations between intervention groups; p = 0.1333, Wilcoxon (Mann-Whitney); Difference in median change = -0.711789 — Estimated value reported as difference in median change from baseline to 4 weeks for the MPFC first group minus the median change from baseline to 4-weeks for the DPFC first group

4. Secondary Outcome: Functional Connectivity Dorsolateral Prefrontal Cortex and Anterior Cingulate Cortex
Description: Functional connectivity of the left dorsolateral prefrontal cortex and left dorsal anterior cingulate cortex measured with fMRI, as defined by the temporal correlation in the blood-oxygen-level-dependent signals of the regions. Higher correlations indicate stronger functional connectivity.
Time Frame: Baseline, 4 weeks
Population: Participants with MRI data for both baseline and after 4 weeks of treatment.
Measure: Mean (Standard Deviation); unit: Pearson correlation (r)
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 2 | 4
Pearson correlation (r)
  Correlation between regions at baseline | -0.0563551 (0.0759435) | 0.0542240 (0.0749761)
  Correlation between regions after 4-week intervention | -0.2974375 (0.2386470) | 0.0960170 (0.1248435)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.1333, Wilcoxon (Mann-Whitney); Exact Wilcoxon rank-sum test of comparing changes in correlations between intervention groups; Difference in median change = 0.2729394 — Reported as difference in median change from baseline to 4 weeks for the MPFC first group minus median change for from baseline to 4-weeks for the DPFC first group

5. Secondary Outcome: Functional Connectivity of the Medial Prefrontal Cortex and Ventral Striatum (Nucleus Accumbens)
Description: Functional connectivity of the left medial prefrontal cortex and ventral striatum (mean of medial prefrontal cortex connectivity to left and right nucleus accumbens) measured with fMRI, as defined by the temporal correlation in the blood-oxygen-level-dependent signals of the regions. Higher correlations indicate stronger functional connectivity.
Time Frame: Baseline, 4 weeks
Population: Participants with MRI data for both baseline and after 4 weeks of treatment.
Measure: Mean (Standard Deviation); unit: Pearson correlation (r)
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 2 | 4
Pearson correlation (r)
  Correlation between regions at baseline | 0.1795790 (0.0957911) | 0.0383048 (0.1329478)
  Correlation between regions after 4-week intervention | -0.0576222 (0.1671134) | 0.0474714 (0.1695334)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.2667, Wilcoxon (Mann-Whitney); Exact Wilcoxon rank-sum test comparing changes in functional connectivity from baseline to 4 weeks between intervention groups; Difference in median change = 0.2676718 — Reported as difference in median change from baseline to 4 weeks for the MPFC first minus the median change from baseline to 4 weeks for the DPFC first group

6. Secondary Outcome: Flanker Inhibitor Control and Attention Test, Age 12+
Description: Summary score of accuracy and reaction time. Higher scores indicate stronger inhibitory control and attention (better ability to attend to relevant stimuli and block out irrelevant stimuli). The reported scores are age-corrected standard scores, which have a population mean of 100 and standard deviation of 15. Means are estimated from mixed models.
Time Frame: Baseline, 4 weeks
Population: Those who had a flanker test at baseline and at 4 weeks (stayed in the study through all TMS treatments).
Measure: Least Squares Mean (Standard Error); unit: age-corrected standard score
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 2 | 3
age-corrected standard score
  Baseline | 115 (6) | 97 (5)
  4 weeks | 106 (6) | 93 (5)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.6829, Mixed Models Analysis — Group by time interaction, with time as second measure date; Mean Difference (Final Values) = 5.0000, Standard Error of Mean 11.0972 — This is the adjusted difference in mean for mPFC first relative to DPFC first

7. Secondary Outcome: Kirby Delay Discounting Questionnaire, 27 Item
Description: Summary score of discounting rate. Scores range from 0.00016 to 0.5, with smaller values indicating a lack of discounting and preference for delayed rewards, and higher values indicating strong discounting and preference for immediate rewards. Higher scores are associated with addictive behaviors. The log of K is reported due to its skewed nature. Values are estimated from a mixed model.
Time Frame: Baseline, 4 weeks
Population: Those with a measure at baseline and 4 weeks.
Measure: Least Squares Mean (Standard Error); unit: Log of overall K
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 2 | 3
Log of overall K
  Baseline | -2.9817 (1.1013) | -3.8350 (0.8992)
  4 weeks | -2.7660 (1.1013) | -3.9792 (0.8992)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.7654, Mixed Models Analysis — Group by time interaction p-value, with time as second (last) measure date; Mean Difference (Final Values) = -0.3599, Standard Error of Mean 1.1018 — This is the adjusted difference in mean for MPFC first relative to DPFC first

8. Secondary Outcome: Number of Days of Stimulant Use in the Past Week (Estimated Change Per Day)
Description: Estimated change per day in number of days of stimulant use in the last week (self-reported) from mixed models. Measured as number of days of methamphetamine use because methamphetamine and other stimulant use were reported separately, and it was not clear if these were on the same or different days. The vast majority of subjects reported using only methamphetamine.
Time Frame: Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks, 8 weeks, 12 weeks
Population: All participants who were randomized/received at least one treatment
Measure: Least Squares Mean (Standard Error); unit: Days of use in last week-change per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Days of use in last week-change per day | -0.1026 (0.04322) | -0.09523 (0.04523)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.9070, Mixed Models Analysis — Group by continuous time interaction; Slope = 0.007388, Standard Error of Mean 0.06256 — Difference in slope for MPFC first versus DPFC first

9. Secondary Outcome: Urine Drug Screen Positive for Stimulant
Description: Urine dipstick positive or not for stimulants (amphetamine, methamphetamine, cocaine)
Time Frame: Baseline, 1 week, 2 weeks, 3 weeks, 4 weeks
Population: All participants who were randomized/received at least one treatment.
Measure: Number (95% Confidence Interval); unit: odds ratio for positive per day in study
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
odds ratio for positive per day in study | 0.8892 [0.7687 to 1.0286] | 0.9921 [0.9770 to 1.0074]
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.1427, GEE logistic regression clustered on ID — Based on group x continuous time interaction in generalized estimating equation logistic regression model clustered on subject. This is like a mixed model but uses empirical standard error estimates that are independent of covariance structure; Odds Ratio, log = 0.1095, 95% CI 2-sided [-0.0369 to 0.2559], Standard Error of Mean 0.0747 — Difference in change in log odds of positive UA for stimulant for MPFC first versus DPFC first. Estimated change in log odds per day in the study

10. Secondary Outcome: Brief Substance Craving Scale (Estimated Change in Score Per Day)
Description: The Brief Substance Craving Scale Score used was the summary score of intensity, frequency and length of cravings in the last 24 hours. Scores based on stimulant craving responses and range from 0-12 with higher scores indicating more craving. Scores are least squared means from mixed models of actual measures, without last observation carried forward or any imputation. Change in score per day estimated from a mixed model.
Time Frame: 12 weeks
Population: Those randomized (who received at least one treatment).
Measure: Least Squares Mean (Standard Error); unit: Estimated change in score per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Estimated change in score per day | -0.04980 (0.02369) | -0.02411 (0.01781)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.3917, Mixed Models Analysis; Slope = 0.02569, Standard Error of Mean 0.02964 — This is the difference in slope for MPFC first relative to DPFC first

11. Secondary Outcome: Brief Addiction Monitor Use Subscale (Estimated Change in Score Per Day)
Description: Use subscale. Scores range from 0 to 12 with higher scores indicating more use. Outcome measures reported as change per day estimated from mixed models.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Population: Those who were randomized and received at least one treatment
Measure: Least Squares Mean (Standard Error); unit: Estimated change in scores per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Estimated change in scores per day | -0.05848 (0.01532) | -0.04089 (0.01204)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.3829, Mixed Models Analysis — Group by continuous time interaction; Slope = 0.01759, Standard Error of Mean 0.01948 — Estimated difference in slope of change per day for MPFC first vs. DLPFC first

12. Secondary Outcome: Brief Addiction Monitor Risk Factors Subscale (Estimated Change in Score Per Day)
Description: Risk factors subscale. Scores range from 0 to 24 with higher scores indicating more risk. Results presented as change in score per day estimated from a mixed model.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Population: Those who were randomized/received at least one treatment
Measure: Least Squares Mean (Standard Error); unit: Estimated change in score per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Estimated change in score per day | -0.1235 (0.04053) | -0.1066 (0.03568)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.7595, Mixed Models Analysis — Group by continuous time interaction; Slope = 0.01691, Standard Error of Mean 0.05400 — Estimated difference in slope of change per day for MPFC first vs. DLPFC first

13. Secondary Outcome: Brief Addiction Monitor Protective Factors Subscale (Estimated Change in Score Per Day)
Description: Protective factors subscale. Scores range from 0 to 24 with higher scores indicating more protection. Change in score per day estimated from mixed model.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Population: Those randomized/received at least one treatment with complete BAM protective factors data at one or more time points
Measure: Least Squares Mean (Standard Error); unit: Estimated change in score per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 4
Estimated change in score per day | -0.00530 (0.03623) | 0.03826 (0.03155)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.3839, Mixed Models Analysis; Slope = 0.04356, Standard Error of Mean 0.04804 — Estimated difference in slope of change per day for MPFC first vs. DLPFC first

14. Secondary Outcome: Brief Addiction Monitor Satisfaction With Progress Toward Achieving Recovery Goals (Estimated Change Per Day)
Description: Item 17, satisfaction with progress toward achieving recovery goals. Scores range from 0 to 4 with higher scores indicating less satisfaction. Reported as change per day estimated from a mixed model.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Population: Those who were randomized/received at least one treatment and had a baseline score for question 17 on the Brief Addiction Monitor.
Measure: Least Squares Mean (Standard Error); unit: Estimated change in score per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Estimated change in score per day | -0.01378 (0.01300) | -0.00833 (0.01003)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.7455, Mixed Models Analysis — Group by continuous time interaction; Slope = 0.005445, Standard Error of Mean 0.01642 — Estimated difference in slope of change per day for MPFC first vs. DLPFC first

15. Secondary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Estimated Change in Score Per Day)
Description: Total score. Scores range from 16 to 80 with higher scores indicating more satisfaction. Scores generally reported as a percent of the maximum possible score, such that scores can be calculated with missing responses as long as less than one-third of responses are missing. This outcome measure is reported as change in score per day estimated from mixed models.
Time Frame: Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks
Population: All those who were randomized/received at least one treatment and had complete baseline data for QLES.
Measure: Least Squares Mean (Standard Error); unit: Estimated change in score per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Estimated change in score per day | 0.003497 (0.09139) | 0.2160 (0.07123)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.0823, Mixed Models Analysis — Group by continuous time interaction; Slope = 0.2125, Standard Error of Mean 0.1159 — Difference in estimated change per day for MPFC first versus DPFC first

16. Secondary Outcome: Patient Health Questionnaire--8 Item Scale (Estimated Change in Score Per Day)
Description: Total score. Scores range from 0 to 24 with higher scores indicating worse depressive symptoms. This outcome measure is reported as change in score per day estimated from mixed models.
Time Frame: Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks
Population: All who were randomized/received at least one treatment
Measure: Least Squares Mean (Standard Error); unit: Estimated change in score per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Estimated change in score per day | -0.08549 (0.05749) | -0.1328 (0.0098)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.5289, Mixed Models Analysis — Group by continuous time interaction; Slope = -0.04735, Standard Error of Mean 0.07382 — Difference in estimated change per day for MPFC first versus DPFC first

17. Secondary Outcome: Generalized Anxiety Disorder 7-item Scale (Estimated Change Per Day)
Description: Total score. Scores range from 0 to 21 with higher scores indicating worse anxiety. This outcome measure is reported as change in score per day estimated from mixed models.
Time Frame: Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks
Population: All participants who were randomized/received at least one treatment
Measure: Least Squares Mean (Standard Error); unit: Estimated change in score per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Estimated change in score per day | -0.05545 (0.05014) | -0.05776 (0.03911)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.9714, Mixed Models Analysis — Group by time interaction; Slope = -0.00231, Standard Error of Mean 0.06359 — Estimated difference in change per day for MPFC first versus DPFC first

18. Secondary Outcome: Assessment of Recovery Capital (Estimated Change Per Day)
Description: Total score. Scores range from 0 to 50 with higher scores indicating greater recovery capital. This outcome measure is reported as change in score per day estimated from mixed models.
Time Frame: Baseline, 4 weeks, 8 weeks, 12 weeks
Population: All participants who were randomized/received at least one treatment.
Measure: Least Squares Mean (Standard Error); unit: Estimated change in score per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Estimated change in score per day | 0.09980 (0.09175) | 0.2266 (0.06983)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.2914, Mixed Models Analysis — Group by continuous time interaction; Slope = 0.1268, Standard Error of Mean 0.1153 — Difference in estimated change per day for MPFC first versus DLPFC first

19. Secondary Outcome: Positive and Negative Affect Scale Positive Affect Score (Estimated Change Per Day)
Description: Positive affect score. Scores range from 10 to 50 with higher scores indicating higher positive affect. Higher positive affect is a better outcome. This outcome measure is reported as change in score per day estimated from mixed models.
Time Frame: Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks
Population: All participants who were randomized/received at least one treatment
Measure: Least Squares Mean (Standard Error); unit: Estimated change in score per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Estimated change in score per day | -0.04983 (0.06358) | 0.1111 (0.04856)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.0573, Mixed Models Analysis — Group by continuous time interaction; Slope = 0.1609, Standard Error of Mean 0.08000 — Difference in estimated change per day for MPFC first versus DPFC first

20. Secondary Outcome: Positive and Negative Affect Scale Negative Affect Score (Estimated Change Per Day)
Description: Negative affect score. Scores range from 10 to 50 with lower scores indicating lower negative affect. Lower negative affect is a better outcome. This outcome measure is reported as change in score per day estimated from mixed models.
Time Frame: Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks
Population: All participants randomized/received at least one treatment who had complete PANAS negative affect data at baseline
Measure: Least Squares Mean (Standard Error); unit: Estimated change in score per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 5 | 5
Estimated change in score per day | -0.08496 (0.06962) | -0.07669 (0.05177)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.9250, Mixed Models Analysis — Group by continuous time interaction; Slope = 0.008267, Standard Error of Mean 0.08675 — Difference in estimated change per day for MPFC first versus DPFC first

21. Secondary Outcome: Pittsburgh Sleep Quality Index (Estimated Change Per Day)
Description: Total score. Scores range from 0 to 21, with lower scores indicating better sleep quality. This outcome measure is reported as change in score per day estimated from mixed models.
Time Frame: Baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks
Population: All who were randomized/received at least one treatment
Measure: Least Squares Mean (Standard Error); unit: Estimated change in score per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Estimated change in score per day | -0.08000 (0.02111) | -0.07924 (0.01649)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.9775, Mixed Models Analysis — Group by continuous time interaction; Slope = 0.000766, Standard Error of Mean 0.02679 — Difference in estimated change per day for MPFC first versus DPFC first

22. Secondary Outcome: Difficulties in Emotion Regulation Scale--Short Form (Estimated Change Per Day)
Description: Total score. Scores range from 18 to 90 with higher values indicating more difficulty with emotional regulation. This outcome measure is reported as change in score per day estimated from mixed models.
Time Frame: Baseline, 4 weeks
Population: All participants who were randomized/received at least one treatment
Measure: Least Squares Mean (Standard Error); unit: Estimated change in score per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Estimated change in score per day | -0.1035 (0.02083) | -0.1010 (0.01416)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.9211, Mixed Models Analysis — Group by continuous time interaction; Slope = 0.002498, Standard Error of Mean 0.02518 — Difference in estimated change per day for MPFC first versus DPFC first

23. Secondary Outcome: UPPS-P Impulsive Behavior Scale, 59-item Revised Version (Estimated Change Per Day)
Description: Summary score. Scores range from 59 to 236 with higher scores indicating more impulsive behavior. This outcome measure is reported as change in score per day estimated from mixed models.
Time Frame: Baseline, 4 weeks
Population: All participants who were randomized/received at least one treatment
Measure: Least Squares Mean (Standard Error); unit: Estimated change in score per day
Arm/Group | DPFC First | MPFC First
Number analyzed (Participants) | 6 | 5
Estimated change in score per day | 0.06023 (0.8642) | -0.2392 (0.2670)
Statistical Analysis 1: Comparison: DPFC First vs MPFC First; Test type: Superiority; p = 0.5269, Mixed Models Analysis — Group by continuous time interaction; Slope = -0.2995, Standard Error of Mean 0.4196 — Difference in estimated change per day for MPFC first versus DPFC first

ADVERSE EVENTS:
Time Frame: 4 weeks, while engaged in TMS treatment.
Description: The only serious adverse event did not arise during a treatment session. It could not be specifically attributed to DPFC stimulation versus MPFC stimulation since participants received both at each treatment session, with groups only differentiated by the order in which they received stimulation within each treatment session.
Arm/Group | DPFC First | MPFC First
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/5
Other Adverse Events (participants affected / at risk) | 4/6 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DPFC First (N=6) | MPFC First (N=5)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) — Participant had chronic suicidal thinking pre-dating TMS treatment. It worsened temporarily while the subject was getting treatment, but the subject did not attribute it to TMS and did wish to not stop treatment because of it.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DPFC First (N=6) | MPFC First (N=5)
Headache (mild) (Nervous system disorders) | 2 (6) | 0 (0)
Pain (Nervous system disorders) | 2 (2) | 0 (0) — Pain during TMS. One participant experienced pain at stimulation site and one experienced pain in ear canal. Considered mild. Resolved immediately or shortly after TMS was completed.
Lightheadedness (Nervous system disorders) | 0 (0) | 1 (1) — Participant felt lightheaded after treatment. Severity was mild. Resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/55/NCT04449055/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/55/NCT04449055/ICF_001.pdf